CLINICAL TRIAL: NCT03457740
Title: Influence of Purity Product Supplements on Muscular Strength, Serum Testosterone Levels, Sexual Function, and Quality of Life
Brief Title: Supplement Study: Strength, Testosterone, Sexual Function, Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Purity Products (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-0038
Record Dates: First submitted 2018-02-22; First posted 2018-03-08 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-02

CONDITIONS: Muscular Weakness; Sexual Behavior; Quality of Life
Keywords: muscular strength; testosterone; sexual function; quality of life
MeSH Terms: conditions — Muscle Weakness; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, placebo controlled, double blind
Who Masked: Participant, Investigator
Masking Description: Double blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formula 1 (Experimental): Formula 1 with nutrients and herbs, 4 capsules daily, 6 weeks
  Interventions: Dietary Supplement: Formula 1
- Formula 2 (Experimental): Formula 2 with nutrients and herbs, 4 capsules daily, 6 weeks
  Interventions: Dietary Supplement: Formula 2
- Placebo (Placebo Comparator): Placebo, 4 capsules daily, 6 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Formula 1 — Dietary supplement for strength, testosterone, sexual function, quality of life
  Arms: Formula 1
Dietary Supplement: Formula 2 — Dietary supplement for strength, testosterone, sexual function, quality of life
  Arms: Formula 2
Dietary Supplement: Placebo — Placebo comparison
  Arms: Placebo

SUMMARY:
Decreased muscle mass (sarcopenia) and strength (dynapenia) are common during aging, with a rate of muscle mass loss that is approximately 6% per decade between 30 and 70 years of age. Muscle mass loss results in reduced strength and physical function (frailty), increased risk for falls and bone fractures, and decreased quality of life. The age-related decrease in testosterone plays a key role in the loss of muscle mass and strength for aging males. There is increasing interest in nutritional and exercise strategies to prevent aging-related losses in muscle mass and strength. Sexual dysfunction has a high prevalence among men (31%), and include erectile difficulties (10%), lack of interest in sex (9%), and inability to achieve orgasm (7%). There are multiple causes including low testosterone. There is growing interest in natural supplements, and this study will compare under double blind procedures two natural supplements with placebo (Men's Perfect Multi Formula and Andro Vitality) that have been formulated by Purity Products. The supplements contain micronutrients, plant extracts, and herbs, with the primary bioactives Rhaponticum carthamoides and magnesium. Rhaponticum carthamoides, commonly known as maral root or Russian leuzea, is a perennial herb that grows in South Siberia, and has been used to enhance muscular and sexual function, but more evidence from properly designed human trials is needed to determine both efficacy and safety. The purpose of this study using a randomized, parallel group design, is to evaluate the effect of two supplements relative to placebo on strength, serum free and total testosterone levels, sexual function, mood state, and quality of life compared to placebo over a 6-week period in 120 males.

DETAILED DESCRIPTION:
STUDY PARTICIPANT RECRUITMENT:

Subjects will be recruited via mass advertising in the Charlotte Metropolitan area. Healthy subjects will be screened during recruitment to determine study eligibility (via email and phone). The Charlotte metropolitan area is the largest in the Carolinas, and the sixth largest metropolitan area in the Southeastern region of the United States. Male participants 40 to 70 years of age will be selected who match the listed inclusion and exclusion criteria (next page). The planned distribution of participants by racial/ethnic groups will reflect the demographics of the metropolitan area [White non-Hispanic (60%), Black non-Hispanic (24%), Hispanic (10%), and Asian or Pacific Islander non-Hispanic (3.5%)]. Those subjects who meet all of the inclusion criteria and none of the exclusion criteria will be enrolled and randomized into the study. The study duration for each subject will be 6 weeks. There will be a total of 3 visits for this study. Following recruitment, there will be a 2-week washout period for PDE5 medications. At each of the three morning visits (7:00-9:00 am), subjects will fill in the symptom log (retrospective 3-week period) and have their blood drawn to analyze serum levels of free and total testosterone, and to be tested for strength (isometric hand grip, leg/lower back, YMCA bench press) and body composition (8-point bioelectrical impedance). All subjects will be required to fast overnight for at least 9 hours prior to each visit. Subjects will also be required to abstain from all vigorous exercise and sexual activity at least 24-hours prior to each visit. Within three days prior to each lab visit, subjects will use Survey Monkey via the Internet to fill in responses to three questionnaires: CSFQ, WHO-QOL, and POMS.

RESEARCH PLAN A. V1 - Baseline Visit - Week 0 Prior to the first lab visit, subjects will be recruited according to the listed inclusion and exclusion criteria. Subjects who agree to participate in the study, will be sent the Informed Consent Document (ICD) for review and signature. Subjects will fill in the Medical Health Questionnaire (MHQ) via Survey Monkey to obtain demographic, lifestyle, and medical histories. Following recruitment, there will be a 2-week washout period for PDE5 medications. Within three days prior to the first lab visit, subjects will supply responses to the CSFQ, WHO-QOL, and POMS Questionnaires via Survey Monkey. The compensation contract will be reviewed and signed.

* Informed Consent: At the first lab visit (V1), all subjects will review the Informed Consent Document (ICD) that was previously sent via email attachment, and receive a signed copy.
* Questionnaires: Responses to the CSFQ, WHO-QOL, and POMS questionnaires sent prior to the first lab visit via Survey Monkey will be reviewed for completeness. Subjects will fill in the symptom log.
* Blood Sample: Subjects will have their blood drawn for analysis of free and total testosterone. Subjects will be asked to come in to the clinic during the early morning having fasted for at least 9 hours prior to the visit and refrained from having sexual intercourse 24 hours prior to the visit.
* Anthropometric and Strength Measures: Subjects will be measured for height and weight, and percent body fat using 8-point BIA. Handgrip and leg/lower back strength will be assessed with dynamometers (Figure 3). Subjects will also be tested for upper body strength using the YMCA bench press test (reps with 80-pound barbell set with a metronome for 30 lifts per minute).
* Randomization and Study Product Dispensing: Subjects will be assigned a randomization number, and receive a 3 week supply of the study product. The study product will be contained in supplement trays with specific dates and instructions applied. Subjects must return the supplement trays at the next two lab visits to verify compliance with the dosing regimen.

B. V2 -Mid-Study Visit (Week 3)

* Retrieval Procedures: Subjects will return their supplement tray and any unused study product.
* Intercurrent Medical History and Concomitant Medication History: Subjects will be interviewed by the clinic staff to determine whether there have been any changes in their medical history, whether they have started taking any new medications.
* Questionnaires: Responses to the CSFQ, WHO-QOL, and POMS questionnaires sent within 3-days prior to the second visit via Survey Monkey will be reviewed for completeness. Subjects will fill in the symptom log (3 week retrospective).
* Blood Sample: Subjects will have their blood drawn for analysis of free and total testosterone. Subjects will be asked to come in to the clinic during the early morning having fasted for at least 9 hours prior to the visit and refrained from having sexual intercourse and all exercise 24 hours prior to the visit.
* Anthropometric and Strength Measures: Subjects will be measured for weight, and percent body fat using 8-point BIA. Handgrip and leg/lower back strength will be assessed with dynamometers, and upper body strength with the YMCA bench press test.
* Study Product Dispensing: Subjects will receive their final 3-week supply of the study supplements. Subjects must return the supplement tray at the final lab visit to verify compliance with the dosing regimen.

C. V3 -End-of-Study Visit (Week 6)

* Retrieval Procedures: Subjects will return their supplement tray and any unused study product.
* Intercurrent Medical History and Concomitant Medication History: Subjects will be interviewed by the clinic staff to determine whether there have been any changes in their medical history, whether they have started taking any new medications.
* Questionnaires: Responses to the CSFQ, WHO-QOL, and POMS questionnaires sent within 3 days prior to the final lab visit via Survey Monkey will be reviewed for completeness. The final symptom log will be completed. The compensation contract will be reviewed.
* Blood Sample: Subjects will have their blood drawn for analysis of free and total testosterone. Subjects will be asked to come in to the clinic during the early morning having fasted for at least 9 hours prior to the visit and refrained from having sexual intercourse 24 hours prior to the visit.
* Anthropometric and Strength Measures: Subjects will be measured for height and weight, and percent body fat using 8-point BIA. Handgrip and leg/lower back strength will be assessed with dynamometers, and upper body strength with the YMCA bench press test.

D. Investigational Study Products Formula 1 - a Men's Perfect Multi Formula boosted by extra Magnesium and key vitamins and co-factors. 4 tablets.

Formula 2 - an Herbal blend - we're naming "AndroVitality" with Rhaponticum, Rhododendron caucasicum, 180 mg magnesium, 10 zinc and 2000 IU vitamin D. 4 tablets.

INSTRUCTIONS: Take 4 capsules daily, with water on an empty stomach. If the study participant reports that they get an upset stomach from ingesting the capsules, they will be allowed to consume a small snack. The investigators will store the study product in a locked cabinet in a limited access room, in accordance with the manufacturer's instructions, i.e. in a dry place and at room temperature. Purity Products will provide the ASU-NCRC Human Performance Lab with sufficient study product to complete this study. The supplements and placebo product, will be supplied to the Primary Investigator (DCN) in boxes using A, B, and C codes so that both the investigators and the subjects will be blinded regarding the type of supplement being ingested. Supplement trays will be given to each subject, and will contain labels with the following information:

* Study code number
* Patient number
* Directions of use
* Storage instructions

E. Concomitant Medication Prohibited Medications and Interventions

The following products and interventions are not permitted while the subject is in this study:

· No erectile dysfunction medications or dietary supplements containing ingredients advertised for influences on sexual function or testosterone.

F. Data Analysis and Statistical Methods Data will be entered into an Excel worksheet under the direction of the Primary Investigator (DCN) and the Research Manager. Data statistical analysis (with identifier information deleted) will be conducted by Drs. Nieman, Canu, and Broman-Fulks. The basic statistical model will be a 3 (group) x 3 (time) repeated measures ANOVA within the SPSS Generalized Linear Model (GLM). Subjects will be randomized in equal numbers to one of three groups: two supplement groups; Placebo. The blinding code will be created by Purity Products and stored in a locked cabinet, and provided to the Primary Investigator AFTER all data have been collected. The file linking ID numbers and names of study participants will be stored at uStor, the secure storage site for Appalachian State University (http://ustorcloud.appstate.edu). Analysis and interpretation of data from the CSFQ, WHO-QOL, and POMS questionnaires will be under the direction of clinical psychologists Drs. Canu and Broman-Fulks. Prior to the initiation of the study, this protocol including the informed consent form will be submitted to the ASU IRB and the trial will not start until unconditional approval is received. All guidelines from the ASU IRB for protection of personal data will be followed. The Primary Investigator will assign a subject number to each subject that will be used for identification whenever subject related data are recorded for the sponsor or reported. Subjects who are randomized, but drop out prior to completing the study will be recorded. A record of reasons why subjects drop out of the study will be maintained. After data analysis the Primary Investigator will summarize the results in a final report which accurately reflects the clinical data of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male, 40 to 70 years of age.
* In a stable relationship during at least the past 3 months, with active sexual relations, and an anticipated stable sexual relationship during the 6-week study period.
* Non-diseased, and in general good health on the basis of medical history.
* Low level of weight lifting in a gym or club setting (history of resistance training less than an average of once per week during the previous 6 months).
* Willingness to maintain current exercise and diet habits during the study.
* No history of a bleeding disorder (e.g., von Willebrand Disease) or current use of medications that affect clotting in the blood.

Exclusion Criteria:

* History of prostate cancer or any physical disability that limits sexual function.
* Receiving any treatment/therapy for sexual disorders during the past 6 months.
* Currently using Viagra, Cialis or Levitra (or similar products), or unwillingness to quit use two weeks prior to the start of the study.
* Currently using dietary supplements with ingredients advertised for their influence on muscle strength, sexual function, or testosterone, or unwillingness to quit use two weeks prior to the start of the study.
* Current personal history of psychiatric illness and/or use of treatment medications.
* Current alcohol and/or drug abuse.
* Current history of bleeding disorder (e.g., von Willebrand Disease) or use of anti-clotting medication.
* Scheduled surgery during the study or within 2 weeks after the study is over.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 118 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Change in leg/back muscle strength | Change from baseline leg/back strength scores at 3 weeks, 6 weeks
  Leg/lower back dynamometer test

SECONDARY OUTCOMES:
Change in serum testosterone | Change from baseline serum testosterone levels at 3 weeks, 6 weeks
  Changes in free and total serum testosterone levels
Change in sexual function | Change from baseline CSFQ scores at 3 weeks, 6 weeks
  Changes in Sexual Functioning Questionnaire (CSFQ) scores
Change in quality of life | Changes from baseline WHO-QOL scores at 3 weeks, 6 weeks
  Changes in World Health Organization Quality of Life (WHO-QOL) scores
Change in mood state | Changes from baseline POMS scores at 3 weeks, 6 weeks
  Changes in Profile of Mood States (POMS) scores
Change in handgrip strength | Changes from baseline handgrip strength scores at 3 weeks, 6 weeks.
  Changes in handgrip dynamometer strength
Change in bench press muscular endurance | Changes from baseline bench press repetitions at 3 weeks, 6 weeks
  Changes in bench press repetitions

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Will depend on journal that publishes the data.